CLINICAL TRIAL: NCT04963621
Title: Child-Adolescent Emotion and Stress Intervention Program for Children With Emotional and Stress Problems- a Randomized Controlled Study
Brief Title: RCT of CESIP for Children With Emotional and Stress Problems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH-20-065
Record Dates: First submitted 2021-07-11; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-03

CONDITIONS: Emotional Stress
Keywords: emotional stress; intervention; RCT
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The evaluator was unaware of the subjects' treatment status
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Child-Adolescent Emotion and Stress Intervention Program
  Interventions: Behavioral: Child-Adolescent Emotion and Stress Intervention Program
- waiting (Active Comparator): treat as usual
  Interventions: Behavioral: Child-Adolescent Emotion and Stress Intervention Program

INTERVENTIONS:
Behavioral: Child-Adolescent Emotion and Stress Intervention Program — Intervention programs include Emotion and Stress Intervention for children with emotional and stress problems

SUMMARY:
To explore the effect of Child-Adolescent Emotion and Stress Intervention Program for children with emotional and stress problems, providing early social psychological intervention for aiming the core impairments of emotional and stress problems.

DETAILED DESCRIPTION:
80 children with emotional and stress problems will be randomly divided into the intervention group and the waiting group. The waiting group received regular clinical intervention, while the intervention group received 12-week training. The intervention program includes emotional regulation and stress intervention training for children by two therapists, which were carried out in one meeting rooms in Xinhua Hospital. Therapists are psychotherapists with a background in child psychotherapy training. After 12 weeks, the improvement of emotional symptoms was compared.

ELIGIBILITY:
Inclusion Criteria:

* The results were positive on the SCARED scale; Age 6 years 0 to 12 years 11 months; Total IQ is above 80 assessed by WPPSI.

Exclusion Criteria:

* Attention deficit disorders resulting from organic neurological diseases, extensive developmental disorders, mental retardation, childhood schizophrenia, mood disorders, epilepsy, and other organic diseases or other primary mental disorders; parent or guardian with a serious mental illness, such as schizophrenia, mood disorder (onset), etc., and Educational level is lower than junior middle school; Participants who failed to attend more than 80% of the intervention sessions (at least 9 sessions).

Ages: 72 Months to 155 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire (SDQ) total score | 12 weeks after baseline
  A strengths and difficulties questionnaire (SDQ) tests behavior by asking questions on 25 different positive and negative attributes.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No